CLINICAL TRIAL: NCT01701557
Title: Fluid Resuscitation for Pediatric Diabetic Ketoacidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0846
Record Dates: First submitted 2012-10-01; First posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes
Keywords: Ketoacidosis Fluids
MeSH Terms: conditions — Diabetes Mellitus | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- slow fluid rate (Active Comparator): bolus 10 ml/kg of NS followed by 1.25 times maintenance rate
  Interventions: Other: slow fluid rate
- Fast fluid rate (Active Comparator): bolus 20 ml/kg of NS followed by 1.5 times maintenance rate
  Interventions: Other: fast fluid rate

INTERVENTIONS:
Other: slow fluid rate — 10 mL/kg of NS intravenous bolus over the first hour followed by ¾ NS with potassium replacement at 1.25 times maintenance
  Other Names: normal saline
  Arms: slow fluid rate
Other: fast fluid rate — 20 mL/kg of NS intravenous bolus over the first hour followed by ¾ NS with potassium replacement at 1.5 times maintenance
  Other Names: normal saline
  Arms: Fast fluid rate

SUMMARY:
Randomized trial to determine if the volume of fluid administration in pediatric patients with DKA impacts the rate of normalization of serum bicarbonate, pH as well as the length of treatment

DETAILED DESCRIPTION:
A randomized trial of two initial volumes of IVF and subsequent administration rates. Group I received 10 mL/kg of NS intravenous bolus over the first hour followed by ¾ NS with potassium replacement at 1.25 times maintenance and Group II received 20 mL/kg of NS intravenous bolus over the first hour followed by ¾ NS with potassium replacement at 1.5 times maintenance. The specific variables measured included demographics (age, gender, and race/ethnicity) and routine laboratory values (pH, pCO2, plasma glucose, electrolytes, bicarbonate, sodium, chloride, BUN. Length of treatment was defined as a time of the hospital stay after the start of IVF infusion.

ELIGIBILITY:
Inclusion Criteria:

* 1 day to 18 years of age
* type 1 diabetes
* presence of DKA, as defined by glucose >250 mg/dl, accumulation of ketone bodies in the blood, and metabolic acidosis (venous pH < 7.30 or serum bicarbonate < 15 mmol/L.)

Exclusion Criteria:

* requirement for additional fluid resuscitation for hemodynamic instability
* weight greater than 70 kilograms

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
time to normalization of bicarbonate and pH | start of treatment until resolution of DKA an expected average of 12 to 24 hours
  Laboratory parameters were measured hourly for the first 4 hours, and every 2 to3 hours thereafter until acid-base normalization (pH was above 7.3 or the HCO3 was above 15 mmol/L)

SECONDARY OUTCOMES:
the length of treatment | discharge from the hospital, an expected average of 1-2 days
  Length of treatment was defined as a time of the hospital stay after the start of IVF infusion

CONTACTS AND LOCATIONS:
Overall Officials: Arleta Rewers, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- the Childrens Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Bakes K, Haukoos JS, Deakyne SJ, Hopkins E, Easter J, McFann K, Brent A, Rewers A. Effect of Volume of Fluid Resuscitation on Metabolic Normalization in Children Presenting in Diabetic Ketoacidosis: A Randomized Controlled Trial. J Emerg Med. 2016 Apr;50(4):551-9. doi: 10.1016/j.jemermed.2015.12.003. Epub 2016 Jan 25. PMID 26823137